CLINICAL TRIAL: NCT02082691
Title: Single Patient IND: Continued Administration of G-202 to a Patient With Advanced Hepatocellular Carcinoma Previously Treated With G-202 and Receiving Clinical Benefit
Brief Title: Continued Administration of G-202 for One Patient With Advanced Hepatocellular Carcinoma
Status: No longer available | Type: Expanded Access
Sponsor: Devalingam Mahalingam (Other)
Collaborators: GenSpera, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Devalingam Mahalingam, Prinicipal Investigator, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Other Study IDs: CTRC 13-0040; HSC20130391T [UTHSCSA IRB]
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: G-202; Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

INTERVENTIONS:
Drug: G-202 — Patient will receive G-202 for 3 days in a row, followed by 25 days without taking G-202. This cycle will be repeated every 28 days. Patient will receive G-202 as long as his/her cancer does not grow and the investigational drug side effects are tolerable.

SUMMARY:
Patient with advanced liver cancer (cancer that has spread to other parts of the body) continues to receive the study drug (G-202) even though patient no longer meets the criteria to be a part of the main treatment study. Patient's cancer responded well to receiving G-202 in the main study and will receive G-202 at the same dose given in the main study.

ELIGIBILITY:
Inclusion Criteria:

* History of hepatocellular carcinoma
* Participation in prior research study where G-202 was administered
* Tolerance of G-202 treatment
* Demonstration of stable disease

Exclusion Criteria:

* Disease progression
* Occurrence of unacceptable toxicity

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Devalingam Mahalingam, MD, Principal Investigator — University of Texas Health Science Center San Antonio